CLINICAL TRIAL: NCT06984679
Title: Comparison of Dyspnea, Functional Capacity, Muscle Strength, Urinary Incontinence and Quality of Life Between Children and Adolescents With Cystic Fibrosis and Healthy Children
Brief Title: Physical Impairments in Children With Cystic Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Healthy and Cystic Fibrosis
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Urinary Incontinence; Dyspnea; Muscle Strength; Quality of Life; Exercise Test
MeSH Terms: conditions — Cystic Fibrosis; Urinary Incontinence; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Group: This group will consist of children and adolescents with cystic fibrosis.
  Interventions: Other: Physical Evaluations in Children with Cystic Fibrosis
- Control Group: This group will consist of healthy children and adolescents.
  Interventions: Other: Physical Evaluations in Healthy Children

INTERVENTIONS:
Other: Physical Evaluations in Children with Cystic Fibrosis — In this study, dyspnea, functional capacity, muscle strength, urinary incontinence and quality of life will be evaluated in children and adolescents with cystic fibrosis. The data to be obtained through all these evaluations will be done face to face within 45-60 minutes.
  Groups: Cystic Fibrosis Group
Other: Physical Evaluations in Healthy Children — In this study, dyspnea, functional capacity, muscle strength, urinary incontinence and quality of life will be evaluated in healthy children and adolescents. The data to be obtained from all these assessments will be made face to face within 45-60 minutes.
  Groups: Control Group

SUMMARY:
It is aimed to reveal impairments regarding urinary incontinence, dyspnea, muscle strength, functional capacity or quality of life in children and adolescents with cystic fibrosis compared to healthy children and adolescents.

DETAILED DESCRIPTION:
This study aims to compare dyspnea, functional capacity, muscle strength, urinary incontinence and quality of life between children and adolescents with cystic fibrosis and healthy children and adolescents. Participants will be assessed for these parameters through clinical evaluations, exercise tests, questionnaires and measurements. The study aims to understand the health implications of cystic fibrosis and provide the basis for improvements in the health management of these individuals.

ELIGIBILITY:
Inclusion Criteria for Children and Adolescents with Cystic Fibrosis:

* To be between the ages of 6-18
* To have been diagnosed with cystic fibrosis
* To be clinically stable for at least 3 weeks
* To have the necessary cooperation for the measurements
* To volunteer to participate in the study

Inclusion Criteria for Healthy Children and Adolescents:

* To be between the ages of 6-18
* To be in a similar average and ratio with the group of children and adolescents with cystic fibrosis in terms of age and gender
* To have the necessary cooperation for the measurements
* To volunteer to participate in the study

Exclusion Criteria for Children and Adolescents with Cystic Fibrosis:

* Having any orthopedic, neurological, psychological or cardiovascular problem that may prevent the measurements from being performed in the last 6 months
* Smoking or quitting smoking

Exclusion Criteria for Healthy Children and Adolescents:

* Having any orthopedic, neurological, psychological or cardiovascular problem that may prevent the measurements from being performed in the last 6 months
* Having any chronic disease
* Smoking or quitting smoking

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: At least 25 patients with cystic fibrosis will be included in the main group and at least 25 healthy individuals will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | through study completion, an average of 1 year
  Grip strength will be measured using a dynamometer. Each hand will be tested three times, and the highest value will be recorded for both sides.

SECONDARY OUTCOMES:
Dyspnea score | through study completion, an average of 1 year
  Dyspnea will be assessed with the Modified Medical Research Council (MMRC) Dyspnea Scale, scored from 0 (no dyspnea) to 4 (maximum severity).
Pulmonary Function Test Evaluation | through study completion, an average of 1 year
  Lung function will be assessed with a spirometer. The highest value of the three measurements will be used and interpreted according to gender, age, weight and height. A value below 80% of the expected value will be interpreted as abnormal.
Respiratory Muscle Strength Evaluation | through study completion, an average of 1 year
  Respiratory muscle strength will be assessed with a spirometer. The test will be conducted with the participant seated, using a mouthpiece and a nose clip. The highest value for inspiratory and expiratory pressure will be recorded. A value below 80% of the expected value will be interpreted as abnormal.
Cough Strength Evaluation | through study completion, an average of 1 year
  The peak cough expiratory flow of the individual will be assessed using a peak flow meter. The best of at least three repetitions is recorded.A value above 450 indicates effective cough.
Aerobic Exercise Capacity Evaluation | through study completion, an average of 1 year
  Aerobic capacity will be assessed twice via 6-minute walk test. The longest distance will be used for analysis. A value below 80% of the expected value will be interpreted as abnormal.
Anaerobic Exercise Capacity Evaluation | through study completion, an average of 1 year
  Anaerobic capacity will be assessed via the 3-minute step test (3-STT). For the 3-STT, participants will rest for 10 minutes before performing the test with a 15 cm step at a rate of 30 steps per minute, controlled by a metronome. The total number of steps will be recorded.A high number of steps indicates good capacity.
Quality of Life Score | through study completion, an average of 1 year
  The scale we will use to assess health-related quality of life, the Pediatric Quality of Life Inventory (PedsQL 4.0). The scale was developed to assess the health-related quality of life of children and adolescents between the ages of 2 and 18 and consists of physical, emotional, social and school functioning items, totaling 23 items.Scores from this questionnaire are converted to a scale of 0 to 100. Higher scores indicate better health-related quality of life.
Urinary incontinence score | through study completion, an average of 1 year
  Urinary incontinence will be assessed using the Voiding Dysfunction Symptom Score, a 15-item questionnaire. A score above 8.5 indicates the presence of lower urinary tract symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, Assoc Prof, Study Director — Izmir Democracy University; Yağmur Külekçi, PT, Principal Investigator — Izmir Democracy University; Gökçen Kartal Öztürk, Assoc Prof, Principal Investigator — Ege University; Ece Ocak, Dr, Principal Investigator — Izmir City Hospital; Kübra Özkaya, Dr, Principal Investigator — Ege University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuğay, B. U., Arıkan, H., & Özçelik, U. (2004). Kistik fibrozisli çocuklarda pulmoner fonksiyonlar ve vücut kompozisyonu ile kas kuvveti arasındaki ilişki. Fizyoterapi ve Rehabilitasyon, 15(2), 47-54.
- [Background] Frayman KB, Kazmerski TM, Sawyer SM. A systematic review of the prevalence and impact of urinary incontinence in cystic fibrosis. Respirology. 2018 Jan;23(1):46-54. doi: 10.1111/resp.13125. Epub 2017 Jul 18. PMID 28718995
- [Background] Heron J, Grzeda MT, von Gontard A, Wright A, Joinson C. Trajectories of urinary incontinence in childhood and bladder and bowel symptoms in adolescence: prospective cohort study. BMJ Open. 2017 Mar 14;7(3):e014238. doi: 10.1136/bmjopen-2016-014238. PMID 28292756